CLINICAL TRIAL: NCT05321537
Title: Comparison of Somatosensory Exercise Versus Endurance-strength Exercise in Patients With Chronic Neck Pain: a Randomized Clinical Trial
Brief Title: Comparison of Somatosensory Versus Endurance-strength Exercise in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexander Achalandabaso (Other)
Responsible Party: Sponsor-Investigator, Alexander Achalandabaso, Clinical professor, University of Jaén
Organization: University of Jaén (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM/2022/1/001
Record Dates: First submitted 2022-03-23; First posted 2022-04-11 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Neck Pain
Keywords: neck pain; chronic pain; therapeutic exercise; proprioception; motor control
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: A single center, parallel, randomized, blinded rater, controlled clinical trial will be conducted. The 25 requirements proposed by the CONSORT declaration will be followed.
Who Masked: Outcomes Assessor
Masking Description: The evaluator will not know to which treatment group each belongs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Somatosensory training (Experimental): It consists of head relocation exercises, eye tracking, gaze stability and eye-head coordination. It requires the use of special material, the pupillary glasses allow the gaze to be fixed by restricting peripheral vision and the laser pointer provides visual feedback on the positioning of the head.
  Interventions: Other: Therapeutic exercises
- Endurance-strength training (Experimental): It consists of low-load training of the craniocervical flexor muscles. This exercise is specific for the deep cervical flexor muscles, while seeking minimal activation of the superficial flexor muscles. This training consists of 5 phases, starting with a pressure of 20 mmHg, progressively increasing 2 mmHg in each phase.
  Interventions: Other: Therapeutic exercises

INTERVENTIONS:
Other: Therapeutic exercises — A somatosensory training and an endurance-strength training protocol

SUMMARY:
Aim: To compare the effects of somatosensory exercise vs endurance-strength exercise on the deep cervical flexor muscles on pain and perceived disability in patients with chronic neck pain.

Study design: Protocol of a clinical trial, controlled, parallel and a blinded assessor.

Population: Subjects aged 18 to 65 years with neck pain of 3 or more months of evolution.

DETAILED DESCRIPTION:
The study will be carried out at the Faculty of Nursing and Physiotherapy of the University of Alcalá. A total of 60 subjects with nonspecific chronic neck pain will be selected and randomly assigned into two intervention groups. The first group will perform a somatosensory exercise program and a second group will perform activation and endurance-strength exercises of the deep cervical flexors. The duration of the intervention will be 8 weeks, with 6 sessions of physical therapy and daily home exercise. The variables pain, pressure pain threshold, disability, endurance-strength, proprioception, quality of life, kinesiophobia, quality of sleep and depression will be analyzed. Measurements will be taken pre-treatment, post-treatment and a follow-up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of age between 18 and 65 years
* Neck pain of 3 or more months of evolution

Exclusion Criteria:

* Cervical Disability Index less than 15/50
* Infection
* Oncological processes
* Neck or arm surgery
* Neck or arm trauma
* Positive neurological signs
* Rheumatic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-19 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Pain change | Pre-intervention, post-intervention (2 months) and follow-up of 3 months after the end.
  To assess pain, the Visual Analogue Scale will be used, which consists of a 10-centimeter horizontal line, at whose ends is the maximum expression of a symptom.
Disability change | Pre-intervention, post-intervention (2 months) and follow-up of 3 months after the end.
  Disability will be assessed using the validated Spanish version of the Cervical Disability Index. Its range score is 0-50, higher values mean greater disability.

SECONDARY OUTCOMES:
Pressure Pain Threshold change | Pre-intervention, post-intervention (2 months) and follow-up of 3 months after the end.
  To assess the Pressure Pain Threshold, a analog pressure algometer will be used. The pressure will be performed bilaterally on the levator scapulae, upper trapezius, splenius capitis and sternocleidomastoid.
Endurance of craniocervical flexion change | Pre-intervention, post-intervention (2 months) and follow-up of 3 months after the end.
  The isometric endurance of the deep flexor muscles of the neck will be measured with the Craniocervical Flexion Test, using a pressure biofeedback.
Proprioception change | Pre-intervention, post-intervention (2 months) and follow-up of 3 months after the end.
  The proprioception of the head and neck in space will be evaluated using the Cervical Joint Positioning Error Test.
Kinesiophobia change | Pre-intervention, post-intervention (2 months) and follow-up of 3 months after the end.
  The patients' level of fear of movement will be evaluated using the Tampa Scale for Kinesiophobia. Range score is 11-44, higher values mean greater fear of injury.
Sleep quality change | Pre-intervention, post-intervention (2 months) and follow-up of 3 months after the end.
  To assess sleep quality we will use the Pittsburgh Sleep Quality Index, using the Spanish version. Range score is 0-21, higher values mean worse outcome.
Quality of life change | Pre-intervention, post-intervention (2 months) and follow-up of 3 months after the end.
  Quality of life will be assessed with the 12-Item Short Form Survey, second version (SF-12v2), using its Spanish version. This questionnaire is made up of 12 items which measure both physical and mental items. Range score is PCS 24-56,6 and MCS 19-60,8, higher values mean higher quality of life.
Depression change | Pre-intervention, post-intervention (2 months) and follow-up of 3 months after the end.
  To assess depression, the Beck Depression Inventory in its second edition (BDI-II), in its Spanish version, will be used. Range score is 0-63, higher values mean worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No